CLINICAL TRIAL: NCT01887639
Title: Prevalence and Risk Factors in Unipolar Depression Patients Without Remission After One Antidepressant Trial: PANTHER Study
Brief Title: Prevalence and Risk Factors in Unipolar Depression Patients Without Remission After One Antidepressant Trial
Acronym: PANTHER
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-NAR-XXX-2013/1
Record Dates: First submitted 2013-06-25; First posted 2013-06-27 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Non-psychotic Unipolar Major Depression
Keywords: Non-psychotic unipolar major depression; Resistant depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Unipolar major depression: Outpatients Individuals between 18 and 75 years old with a current episode of non-psychotic unipolar major depression that are treated with an antidepressant drug according to physician´s current and usual practice.

SUMMARY:
A non interventional, descriptive, longitudinal cohort study is designed, trying to obtain local data about the prevalence of non remitted depressed patients after an antidepressant treatment, and to get information about sociodemographic and clinical characteristics of these patients as well as features of their treatments and compare them with those of the patients that achieve remission. Also the effect of patient´s expectation in the treatment outcome will be examined.

DETAILED DESCRIPTION:
A non interventional, descriptive, longitudinal cohort study is designed, trying to obtain local data about the prevalence of non remitted depressed patients after an antidepressant treatment, and to get information about sociodemographic and clinical characteristics of these patients as well as features of their treatments and compare them with those of the patients that achieve remission. Also the effect of patient´s expectation in the treatment outcome will be examined.

Non psychotic depressed patients that are initiating an antidepressant treatment will be recruited. Socio demographic and clinical features will be recorded as well as their expectations before the treatment. Severity of depression and treatment characteristics will be recorded after 4 to 8 weeks of drug treatment at an adequate dose. Variables will be compared between the patients that will achieve remission and those that do not.

ELIGIBILITY:
Inclusion Criteria:

Female and male aged 18 to 75 years old. Outpatients with a current episode of non-psychotic unipolar major depression according to the DSM IV-TR.

Severity of illness assessed by means of a score ≥ 14 in the HAM D17 Have not been medicated for the current depression episode with an antidepressant Provision of subject informed consent

Exclusion Criteria:

Patients participating in any clinical trial, the subject cannot take part in this study.

The individual has participated in the last 3 months (including this study) or is participating in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals between 18 and 75 years old that have non-psychotic unipolar major depression and have not been treated for the current episode.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with unipolar major depression that do not achieve remission after one antidepressant treatment. | 12 weeks
  Non psychotic depressed patients that are initiating an antidepressant treatment will be recruited. Socio demographic and clinical features will be recorded as well as their expectations before the treatment. Severity of depression and treatment characteristics will be recorded after drug treatment at an adequate dose. Variables will be compared between the patients that will achieve remission and those that do not.

SECONDARY OUTCOMES:
Clinical, therapeutic and socio-demographic characteristics of resistant depression patients and comparisson of them with the characteristics of the sample of depressed patients in remission. | 12 weeks
  Description of the clinical (Clinical history, episode features, BDI and HAM D17 scores), therapeutic (Type of drug, dose used, treatment period, adherence, presence and type of psychosocial therapy) and socio-demographic (age, gender, civil status, employment status, cohabitation, health insurance) characteristics of resistant depression patients and to compare them with the characteristics of the sample of depressed patients in remission.
Comparison of the depression severity change assessed by the physician with the evaluation done by the patient | 12 weeks
  Comparison of the depression severity change assessed by the physician with the evaluation done by the patient by means of the BDI.

CONTACTS AND LOCATIONS:
Locations (8):
- Argentina (8):
  - Research Site, Buenos Aires
  - Research Site, Caba
  - Research Site, Chaco
  - Research Site, Córdoba
  - Research Site, Rosario
  - Research Site, San Miguel de Tucumán
  - Research Site, San Salvador de Jujuy
  - Research Site, Santa Fe

REFERENCES:
- See also: Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1832&filename=NIS-NAR-XXX-2013-1_AZ_Synopsis.pdf